CLINICAL TRIAL: NCT04179292
Title: The Effect of Physiotherapy Program in Scleroderma Patients: A Randomized Clinical Trial
Brief Title: The Effect of Physiotherapy Program in Scleroderma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Tugba Civi Karaaslan, Research Assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IstanbulU2
Record Dates: First submitted 2019-11-06; First posted 2019-11-27 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Scleroderma; Systemic Sclerosis; Hand Rheumatism; Physiotherapy; Rehabilitation
Keywords: Scleroderma; Systemic sclerosis; Hand therapy
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Systemic | interventions — Physical Therapy Modalities; Rehabilitation

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiotherapy Program (Experimental): Stretching and strengthening exercises, functional exercises, massage techniques, sensory training and breathing exercises will be applied to the patients by physiotherapist for 3 sessions per week. On the other days, it will be implemented as an 8-week home program with 5 sessions per week.
  Interventions: Other: Hand Therapy by Physiotherapist
- Home Program (Experimental): Stretching and strengthening exercises, functional exercises, massage techniques, sensory training and breathing exercises will be applied to the patients as home program. Motivation will be provided by contacting by phone / call once a week for follow-up.
  Interventions: Other: Hand Therapy as home program

INTERVENTIONS:
Other: Hand Therapy by Physiotherapist — stretching exercises; all finger joints, wrist and supination-pronation direction strengthening exercises; finger and wrist functional exercises retrograde massage; starting from the distal phalanx to the elbow sensory education; desentilation training (cotton…) breathing exercises 5 days / week, 8 weeks in total
  * 3 days / week with physiotherapist
  * 2 days / week as home program 30 minutes / day 12 repetitions
  Other Names: Physiotherapy and Rehabilitation
  Arms: Physiotherapy Program
Other: Hand Therapy as home program — stretching exercises; all finger joints, wrist and supination-pronation direction strengthening exercises; finger and wrist functional exercises retrograde massage; starting from the distal phalanx to the elbow sensory education; desentilation training (cotton…) breathing exercises 5 days / week, 8 weeks in total
  * 3 days / week with physiotherapist
  * 2 days / week as home program 30 minutes / day 12 repetitions
  Other Names: Physiotherapy and Rehabilitation
  Arms: Home Program

SUMMARY:
The aim of this study was to investigate the effectiveness of physiotherapy and rehabilitation program on hand involvement of patients with scleroderma and to compare the effects of home rehabilitation program and rehabilitation program under physiotherapist supervision. At the end of the study, the rehabilitation program under the supervision of physiotherapist and home exercise program will be compared with the effects of these applications on range of motion, grip strength, function and sensation. Since there are a limited number of randomized controlled studies in the literature on this subject and there is no randomized controlled clinical study on the superiority of physiotherapist supervision and home program, it will contribute to the information regarding the rehabilitation of scleroderma patients.

DETAILED DESCRIPTION:
Scleroderma is an autoimmune connective tissue disease with fibrosis. Although its etiology and pathogenesis have not been clearly defined, it has a chronic course. It is estimated that scleroderma affects approximately 300,000 people in the United States. Most commonly, it affects adults and women.

When the current literature is examined, Landim et al. in their studies for the development and evaluation of hand exercises home program in patients with systemic scleroderma; They found that the 8-week home exercise program had positive effects on pain, function, mobility and strength. Antonioli et al. concluded that individualized rehabilitation program could improve quality of life and hand mobility in patients with systemic sclerosis. Lopes et al. found that the degree of physical disability was related to both hand grip strength and pulmonary function, but there was no relationship between hand grip strength and pulmonary function in these patients. Mancuso et al. In their case series studies examining the effect of paraffin and exercise on hand functions in scleroderma, they concluded that paraffin and hand exercises can be used to improve hand functions related to participation in daily activities. Rannou et al. in their study comparing the effects of physical therapy program and the usual care of patients with systemic sclerosis on disability, they concluded that 1-month individualized supervised physical therapy program followed by home exercise programs provided short-term benefit. Bongi et al. systemic scleroderma patients with general rehabilitation programs applied to the hand and face specific programs designed to evaluate the effectiveness of their studies; have shown that these techniques improve disability, HRQoL, hand and face functionality.

A limited number of studies in the literature emphasize the need for more research with larger sample size and more variable control.

The aim of this study was to investigate the effectiveness of physiotherapy and rehabilitation program on hand affected patients with scleroderma diagnosis and to compare the effects of home exercise program with physiotherapist supervision. At the end of the study, the rehabilitation program under the supervision of physiotherapist will be compared with the home exercise program and data on the effects of these applications on range of motion, grip strength, function and sensation will be obtained; their superiority to each other will be revealed.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with scleroderma
* Stability of medical treatments
* To be able to adapt to the exercises

Exclusion Criteria:

* The patient has a history of neurological disease or trauma that may affect his symptoms
* Systemic involvement that affects the treatment process
* Being in the active phase of the disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2020-11-21 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
Hand Mobility in Scleroderma (HAMIS) | before treatment, at 8 weeks, 16 weeks, and 12 months change
  Hand Mobility in Scleroderma is a hand function test developed for adults who have systemic sclerosis. HAMIS consists of 9 items designed to measure all movements assessed in an ordinary range of motion-measured hand test. Each item is graded on a 0-3 scale, where 0 corresponds to normal function and 3 denotes that the individual is unable to perform the item. Each hand is assessed separately. The total score of HAMIS for each hand is 370 Sandqvist and Eklund Vol. 13, No. 6, December 2000 27, which represents a high degree of dysfunction.

SECONDARY OUTCOMES:
9-Hole Peg Test | before treatment, at 8 weeks, 16 weeks, and 12 months change
  It is used to evaluate patients' hand and finger skills. The pegboard is placed in the middle of the body. It is desirable that 9 wooden pins be placed randomly in the 9-hole wooden block as fast as possible, and then the pins are removed from the wooden block and placed in the storage compartment one by one. These times are measured and recorded with a stopwatch. A total of 20 seconds or more is considered a "loss of skill".
Duruöz Hand Index | before treatment, at 8 weeks, 16 weeks, and 12 months change
  The Duruoz Hand Index (DHI) is a self-report questionnaire designed to evaluate activity limitations of the hand. This scale contains 18 items. Every item has a score between 0-5 and total score changes between 0-90. Higher scores indicate severe hand-related disability.
Scleroderma Health Assessment Questionnaire (SHAQ) | before treatment, at 8 weeks, 16 weeks, and 12 months change
  The Scleroderma Health Assessment Questionnaire is a measurement tool for evaluating function in individuals with systemic scleroderma and has been used in a number of countries. SHAQ is made up of 20 items distributed among eight domains and has five additional domains that assess dysfunctions caused by the symptoms of systemic scleroderma. For this, five visual analogue scales (VASs) are used. The scores on these scales are converted to subscores ranging from 0 to 3 points. The overall score of the questionnaire is the sum of each of the five VAS subscores and the scores for the eight domains, divided by 13. Lower score indicates better health status.
Semmes Weinstein Monofilaman Test | before treatment, at 8 weeks, 16 weeks, and 12 months change
  The severity of pain and paresthesia symptoms of the patients will be assessed using the 10 cm Visual Analogue Scale. Before the assessment, patients instruct that "0" for "no symptoms", "10" represents "the most severe pain that could be felt" and should mark the point that best describes the symptom. The patient's rest, activity and night pain in the last week will be questioned separately. To evaluate the paresthesia, the most severe paresthesia felt by the patient in the last 1 week will be questioned and it will be asked to mark the place that best expresses paresthesia on the scale. Marked points measure by a ruler and record in centimeters.
Pittsburgh Sleep Quality Index (PSQI) | before treatment, at 8 weeks, 16 weeks, and 12 months change
  The Pittsburgh Sleep Quality Index is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score. Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Fatigue Severity Scale (FSS) | before treatment, at 8 weeks, 16 weeks, and 12 months change
  The Fatigue Severity Scale is a 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders. Answers are scored on a seven point scale where 1 = strongly disagree and 7 = strongly agree. This means the minimum score possible is nine and the highest is 63. The higher the score, the more severe the fatigue is and the more it affects the person's activities.

CONTACTS AND LOCATIONS:
Overall Officials: TUGBA CIVI KARAASLAN, MSc, Principal Investigator — Research Assistant
Locations (1):
- Tugba Civi Karaaslan, Istanbul, Buyukcekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Distler O, Cozzio A. Systemic sclerosis and localized scleroderma--current concepts and novel targets for therapy. Semin Immunopathol. 2016 Jan;38(1):87-95. doi: 10.1007/s00281-015-0551-z. Epub 2015 Nov 17. PMID 26577237
- [Background] Vehe RK, Riskalla MM. Collagen Vascular Diseases: SLE, Dermatomyositis, Scleroderma, and MCTD. Pediatr Rev. 2018 Oct;39(10):501-515. doi: 10.1542/pir.2017-0262. No abstract available. PMID 30275033
- [Background] Landim SF, Bertolo MB, Marcatto de Abreu MF, Del Rio AP, Mazon CC, Marques-Neto JF, Poole JL, de Paiva Magalhaes E. The evaluation of a home-based program for hands in patients with systemic sclerosis. J Hand Ther. 2019 Jul-Sep;32(3):313-321. doi: 10.1016/j.jht.2017.10.013. Epub 2017 Dec 1. PMID 29198478
- [Background] Antonioli CM, Bua G, Frige A, Prandini K, Radici S, Scarsi M, Danieli E, Malvicini A, Airo P. An individualized rehabilitation program in patients with systemic sclerosis may improve quality of life and hand mobility. Clin Rheumatol. 2009 Feb;28(2):159-65. doi: 10.1007/s10067-008-1006-x. Epub 2008 Sep 16. PMID 18795394
- [Background] Lopes AJ, Justo AC, Ferreira AS, Guimaraes FS. Systemic sclerosis: Association between physical function, handgrip strength and pulmonary function. J Bodyw Mov Ther. 2017 Oct;21(4):972-977. doi: 10.1016/j.jbmt.2017.03.018. Epub 2017 Mar 29. PMID 29037654
- [Background] Mancuso T, Poole JL. The effect of paraffin and exercise on hand function in persons with scleroderma: a series of single case studies. J Hand Ther. 2009 Jan-Mar;22(1):71-7; quiz 78. doi: 10.1016/j.jht.2008.06.009. Epub 2008 Aug 30. PMID 18950987
- [Background] Rannou F, Boutron I, Mouthon L, Sanchez K, Tiffreau V, Hachulla E, Thoumie P, Cabane J, Chatelus E, Sibilia J, Roren A, Berezne A, Baron G, Porcher R, Guillevin L, Ravaud P, Poiraudeau S. Personalized Physical Therapy Versus Usual Care for Patients With Systemic Sclerosis: A Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2017 Jul;69(7):1050-1059. doi: 10.1002/acr.23098. Epub 2017 Jun 7. PMID 27696703
- [Background] Schapira AH, Holt IJ, Sweeney M, Harding AE, Jenner P, Marsden CD. Mitochondrial DNA analysis in Parkinson's disease. Mov Disord. 1990;5(4):294-7. doi: 10.1002/mds.870050406. PMID 1979656